CLINICAL TRIAL: NCT07377448
Title: Respiratory Muscle Strength, Pulmonary Function, and Post-Exercise Recovery Responses According to Insulin Use in Individuals With Type 2 Diabetes Mellitus
Brief Title: Insulin Use and Respiratory Muscle Strength in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, Assistant Professor, Izmir Bakircay University
Other Study IDs: 2468
Record Dates: First submitted 2026-01-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 2 Treated With Insulin
Keywords: Insulin Therapy; Respiratory Muscle Strength; Maximal Inspiratory Pressure; Maximal Expiratory Pressure; Spirometry
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Insulin-Treated Type 2 Diabetes Mellitus: Participants with type 2 diabetes mellitus who are currently using insulin therapy as part of usual care at the time of assessment.
- Non-Insulin-Treated Type 2 Diabetes Mellitus: Participants with type 2 diabetes mellitus who are not using insulin therapy as part of usual care at the time of assessment (e.g., lifestyle and/or oral antidiabetic agents).

SUMMARY:
This study compares breathing function, breathing muscle strength, and recovery after a walking test in adults with type 2 diabetes, based on whether they use insulin.

People with type 2 diabetes will be evaluated during a single study visit at Izmir Bakircay University. Participants will be grouped as either currently using insulin or not using insulin as part of their usual diabetes treatment. All participants will complete the same tests: a breathing test (spirometry), breathing muscle strength tests (maximal inspiratory and expiratory pressures), and a 6-minute walk test.

Before the walk test, immediately after the test, and 5 minutes after the test, recovery measures such as heart rate, oxygen saturation, blood pressure, and perceived shortness of breath and fatigue will be recorded. The goal is to understand whether insulin use is associated with differences in breathing and recovery responses in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70 years
* Diagnosis of type 2 diabetes mellitus for at least 1 year
* Receiving diabetes treatment (oral antidiabetic agents and/or insulin) for at least 6 months
* Stable metabolic status (HbA1c ≤ 10%)
* Independent ambulation
* Able to read and understand Turkish
* Provided written informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Active diabetic foot ulcer
* Acute respiratory tract infection or known chronic respiratory disease (e.g., COPD, asthma, interstitial lung disease)
* Cardiovascular disease history that may limit exercise testing (e.g., heart failure, uncontrolled hypertension, arrhythmia)
* Neurological disease, musculoskeletal problem, or balance disorder precluding participation in the exercise test
* Major surgery within the past 6 months
* Current cancer treatment or history of malignancy
* Cognitive impairment or psychiatric condition limiting cooperation
* Pregnancy or breastfeeding

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 40-70 years with a diagnosis of type 2 diabetes mellitus who attended the Izmir Bakircay University Physiotherapy and Rehabilitation Research and Practice Center and met the eligibility criteria. Participants were categorized as insulin-treated or non-insulin-treated based on current usual care.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Single Visit (Baseline)
  Maximal inspiratory pressure (cmH2O) assessed using a respiratory pressure meter according to standardized respiratory muscle strength testing procedures. The best value from repeated acceptable maneuvers will be used for analysis.

SECONDARY OUTCOMES:
Maximal Expiratory Pressure (MEP) | single Visit (Baseline)
  Maximal expiratory pressure (cmH2O) assessed using a respiratory pressure meter. The best value from repeated acceptable maneuvers will be used.
Spirometry Parameters (FVC) Forced Vital Capacity | Single Visit (Baseline)
  Pulmonary function measured by spirometry following standard procedures.
6-Minute Walk Distance (6MWD) | Single Visit (During 6-Minute Walk Test)
  Total distance walked in 6 minutes (meters) on a standardized 30-meter corridor using standardized instructions.
Heart Rate Response and Recovery After the 6-Minute Walk Test | Pre-Test; Immediately Post-Test; 5 Minutes Post-Test
  Heart rate (beats/min) recorded at the specified time points using pulse oximetry.
Oxygen Saturation (SpO₂) Response and Recovery After the 6-Minute Walk Test | Pre-Test; Immediately Post-Test; 5 Minutes Post-Test
  Peripheral oxygen saturation (SpO₂, %) recorded at the specified time points using pulse oximetry.
Blood Pressure Response and Recovery After the 6-Minute Walk Test | Pre-Test; Immediately Post-Test; 5 Minutes Post-Test
  Systolic and diastolic blood pressure (mmHg) measured in a seated position at the specified time points.
Forced Expiratory Volume in 1 Second (FEV1) | Single Visit (Baseline)
  Pulmonary function measured by spirometry following standard procedures.
FEV1/FVC Ratio | Single Visit (Baseline)
  Calculated from spirometry values following standard procedures.
Peak Expiratory Flow (PEF) | Single Visit (Baseline)
  Pulmonary function measured by spirometry following standard procedures.
Rating of Perceived Dyspnea During Recovery (Modified Borg Dyspnea Scale, 0-10) | Pre-Test; Immediately Post-Test; 5 Minutes Post-Test
  Perceived dyspnea will be assessed using the Modified Borg Dyspnea Scale (0 = no breathlessness at all; 10 = maximal breathlessness). Higher scores indicate worse dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakircay University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared